CLINICAL TRIAL: NCT04824300
Title: The Effect of Erector Spina Plane Block on Postoperative Pain and Opiod Consumption After Mastectomy
Brief Title: Efect of Erector Spina Plane Block on Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Meliha Orhon, assistant professor, Marmara University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 09.2020.125
Record Dates: First submitted 2021-03-27; First posted 2021-04-01 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Pain, Postoperative; Opioid Use
Keywords: erector spinae plane block; opioid consumption; mastectomy; Analgesia nosiseption index
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- erector spinae plane block group (Active Comparator): All patients were monitored with standard monitoring (electrocardiography (ECG), noninvasive blood pressure, peripheral oxygen saturation (SpO2)), bispectral index (BIS, Medtronic, Mineapolis) and ANI (analgesia nociception index) -90-120 min) data were recorded.Group ESPB was applied before general anesthesia by the same anesthesiologist with block experience. In the sitting position, using an ultrasound-guided linear probe (6-13 MHz) on the side to be operated, T3 is marked 3 cm from the lateral of the spinous processes and with the in-plane technique, a 22G block needle (100mm, B-Braun, Germany) in the cranio-caudal direction first After it was observed that the erector spina muscle was separated from the transverse process with -2 ml normal saline, 20 ml 0.5% bupivacaine and 100 mg lidocaine were administered. And the drug was found to spread to the craniocaudal line at the ESP on ultrasound.Postoperative pain of the patients was evaluated using VAS (visual analogue scale).
  Interventions: Procedure: erector spinae block
- non block control group (No Intervention): All patients were monitored with standard monitoring (electrocardiography (ECG), noninvasive blood pressure, peripheral oxygen saturation (SpO2)), bispectral index (BIS, Medtronic, Mineapolis) and ANI (analgesia nociception index) -90-120 min) data were recorded.15 minutes before the end of the surgery, 1 gr paracetamol and 100 mg tramadol were given to the control group. Postoperative pain of the patients was evaluated using VAS (visual analogue scale).

INTERVENTIONS:
Procedure: erector spinae block — Erector spina plane block (ESP) is a technique used in many surgeries for anesthesia and analgesia. It is frequently preferred by anesthesiologists for postoperative analgesia recently because it is easy to apply and no complications are reported in the literature. Erector spina muscle, with arms of iliocostalis, longissimus and spinalis, is located parallel to the spine, from the back of the skull to the pelvis. The injected local anesthetic is distributed in many levels in the cranio-caudal direction and blocks the intercostal spinal nerves, causing sensory block. Providing the necessary perioperative analgesia due to the complex innervation of the breast tissue is a big controversy among anesthesiologists. Multimodal analgesia methods with various regional blocks are more preferred. Erector Spina Plane block is also preferred as another method since it provides both perioperative and postoperative analgesia
  Arms: erector spinae plane block group

SUMMARY:
After breast cancer surgery, more than 60% of patients experience persistent pain.Although opioids are the main method of use in postoperative pain management, there are side effects such as constipation, sedation, respiratory depression, urinary retention, itching, postoperative nausea and vomiting.Erector spina plane block (ESPB) is a technique used in many surgeries for anesthesia and analgesia.It is frequently preferred by anesthesiologists for postoperative analgesia recently because it is easy to apply and no complications are reported in the literature.ESPB with arms of iliocostalis, longissimus and spinalis, is located parallel to the spine, from the back of the skull to the pelvis.The injected local anesthetic is distributed in many levels in the cranio-caudal direction and blocks the intercostal spinal nerves, causing sensory block.Providing the necessary perioperative analgesia due to the complex innervation of the breast tissue is a big controversy among anesthesiologists.Multimodal analgesia methods with various regional blocks are more preferred.ESPB block is also preferred as another method since it provides both perioperative and postoperative analgesia.In studies conducted on cadavers, it has been shown that local analgesia spreads to the paravertebral area when applied under the Erektor Spina muscle.Technically, compared to the paravertebral block,the ESPB has proven to be more reliable and easier in terms of pleural puncture risk.

ANI is a monitoring method used in the evaluation of acute nociception and pain.Analyzes the instantaneous changes in heart rate due to the activation of the parasympathetic nervous system using respiratory sinus arrhythmia.A value between 0-100 is obtained.If parasympathetic modulation is very low, a value of 0 is obtained, if it is high, a value of 100 is obtained.ANI detects the noxious stimulus more specifically and sensitively than heart rate and blood pressure changes.

Application of anesthesia and having ANI value between 50-70 in the early postoperative period indicates that analgesia is sufficient,and values <50 are the following 10 minutes.Hemodynamic reactivity (20% increase in heart rate or blood pressure) will occur and the level of analgesia is insufficient,and values> 70 indicate that there is no painful stimulus or that more analgesic drugs are used.

DETAILED DESCRIPTION:
After breast cancer surgery, more than 60% of patients experience persistent pain (1). Although opioids are the main method of use in postoperative pain management, there are side effects such as constipation, sedation, respiratory depression, urinary retention, itching, postoperative nausea and vomiting (2). Erector spina plane block (ESP) is a technique used in many surgeries for anesthesia and analgesia. It is frequently preferred by anesthesiologists for postoperative analgesia recently because it is easy to apply and no complications are reported in the literature. Erector spina muscle, with arms of iliocostalis, longissimus and spinalis, is located parallel to the spine, from the back of the skull to the pelvis. The injected local anesthetic is distributed in many levels in the cranio-caudal direction and blocks the intercostal spinal nerves, causing sensory block (3). Providing the necessary perioperative analgesia due to the complex innervation of the breast tissue is a big controversy among anesthesiologists. Multimodal analgesia methods with various regional blocks are more preferred. Erector Spina Plane block is also preferred as another method since it provides both perioperative and postoperative analgesia (4). In studies conducted on cadavers, it has been shown that local analgesia spreads to the paravertebral area when applied under the Erektor Spina muscle. Technically, compared to the paravertebral block, the Erektor Spina block has proven to be more reliable and easier in terms of pleural puncture risk (5).

ANI is a monitoring method used in the evaluation of acute nociception and pain (Figure 2.1). Analyzes the instantaneous changes in heart rate due to the activation of the parasympathetic nervous system using respiratory sinus arrhythmia. A value between 0-100 is obtained. If parasympathetic modulation (stress level eg presence of pain) is very low, a value of 0 is obtained, if it is high, a value of 100 is obtained (7). ANI detects the noxious stimulus more specifically and sensitively than heart rate and blood pressure changes (6).

The "yellow colored value" on the upper right corner of the ANI monitor shows the instantaneous ANI value, while the orange colored one shows the average ANI value in the last 4 minutes. (Figure 2.1). Application of anesthesia and having ANI value between 50-70 in the early postoperative period indicates that analgesia is sufficient, and values <50 are the following 10 minutes. A hemodynamic reactivity (20% increase in heart rate or blood pressure) will occur and the level of analgesia is insufficient, and values> 70 indicate that there is no painful stimulus or that more analgesic drugs are used (6). After breast cancer surgery, more than 60% of patients experience persistent pain (1). Although opioids are the main method of use in postoperative pain management, there are side effects such as constipation, sedation, respiratory depression, urinary retention, itching, postoperative nausea and vomiting (2). Erector spina plane block (ESP) is a technique used in many surgeries for anesthesia and analgesia. It is frequently preferred by anesthesiologists for postoperative analgesia recently because it is easy to apply and no complications are reported in the literature. Erector spina muscle, with arms of iliocostalis, longissimus and spinalis, is located parallel to the spine, from the back of the skull to the pelvis. The injected local anesthetic is distributed in many levels in the cranio-caudal direction and blocks the intercostal spinal nerves, causing sensory block (3). Providing the necessary perioperative analgesia due to the complex innervation of the breast tissue is a big controversy among anesthesiologists. Multimodal analgesia methods with various regional blocks are more preferred. Erector Spina Plane block is also preferred as another method since it provides both perioperative and postoperative analgesia (4). In studies conducted on cadavers, it has been shown that local analgesia spreads to the paravertebral area when applied under the Erektor Spina muscle. Technically, compared to the paravertebral block, the Erektor Spina block has proven to be more reliable and easier in terms of pleural puncture risk (5).

ANI is a monitoring method used in the evaluation of acute nociception and pain (Figure 2.1). Analyzes the instantaneous changes in heart rate due to the activation of the parasympathetic nervous system using respiratory sinus arrhythmia. A value between 0-100 is obtained. If parasympathetic modulation (stress level eg presence of pain) is very low, a value of 0 is obtained, if it is high, a value of 100 is obtained (7). ANI detects the noxious stimulus more specifically and sensitively than heart rate and blood pressure changes (6).

The "yellow colored value" on the upper right corner of the ANI monitor shows the instantaneous ANI value, while the orange colored one shows the average ANI value in the last 4 minutes. (Figure 2.1). Application of anesthesia and having ANI value between 50-70 in the early postoperative period indicates that analgesia is sufficient, and values <50 are the following 10 minutes. A hemodynamic reactivity (20% increase in heart rate or blood pressure) will occur and the level of analgesia is insufficient, and values> 70 indicate that there is no painful stimulus or that more analgesic drugs are used (6).

ELIGIBILITY:
Inclusion Criteria:

adult female patients ASA 1-3 25-70 years old were included in the study.

Exclusion Criteria:

Severe respiratory and heart disease liver or kidney failure coagulopathy local infection at the injection site spine or chest wall deformity allergy to drugs to be used opioid addiction

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
intraoperative opioid consumption | during surgery
  measurement with analgesia nosiception index monitor

SECONDARY OUTCOMES:
postoperative changes in vas ( visual analog scor) | postoperative first 24 hours.
  recorde postoperative vas changes by anesthesist

CONTACTS AND LOCATIONS:
Overall Officials: MELIHA ORHON ERGUN, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)